CLINICAL TRIAL: NCT06797167
Title: A POST-MARKET, CONFIRMATORY, INTERVENTIONAL CLINICAL INVESTIGATION to EVALUATE the PERFORMANCE and SAFETY of VAGINAL FILLER for the CORRECTION of ATROPHY of the FEMALE EXTERNAL GENITAL AREAS (LABIA MAJORA), RE-PROPORTIONING the RATIO BETWEEN LABIA MINORA and LABIA MAJORA and AMELIORATING SEXUAL FUNCTIONS.
Brief Title: POST-MARKETING CLINICAL STUDY to EVALUATE the EFFICACY and SAFETY of the VAGINAL FILLER MEDICAL DEVICE in CORRECTING THINNING of the GENITAL TISSUE of the LABIA MAJORA in WOMEN, RE-PROPORTIONING the FEMALE EXTERNAL GENITAL AREA and IMPROVING SEXUAL FUNCTION.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rose Pharma SA (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-VAGIFIL-2021
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Atrophy Vulva

STUDY DESIGN:
Intervention Model Description: 76 subjects are enrolled and randomly assigned to one of the two arms with a 1:1 ratio.
  38 subjects will receive the investigational product Vaginal Filler according to the Instruction For Use (IFU); the control group will consist of 38 untreated subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Vaginal Filler) (Experimental): Considering a drop out rate of 10%, 76 female subjects (38 patients per group) will be enrolled. Subjects will be randomly assigned to one of the two arms with a 1:1 ratio: 38 subjects will receive the investigational product, the control group will consist of 38 untreated subjects.
  If assigned to the Vaginal Filler treatment group, participants will be administered the Vaginal Filler device via microinjections into the labia majora.
  Vaginal Filler is a resorbable medical device (physiological, apyrogenic, sterile gel) to be used as a filler to correct hypotrophy, improve the shape and increase the volume of the female external genital areas (labia majora). The main component is cross-linked hyaluronic acid of non-animal origin, produced by bacterial fermentation cross-linked with 1,4-butanediol diglycidyl ether (BDDE).
  Interventions: Device: Injections of a filler gel containing cross-linked hyaluronic acid
- Control Group (No Intervention): Considering a drop out rate of 10%, 76 female subjects (38 patients per group) will be enrolled. Subjects will be randomly assigned to one of the two arms with a 1:1 ratio: 38 subjects will receive the investigational product, the control group will consist of 38 untreated subjects.
  Researchers will compare subjects treated with Vaginal Filler medical device to untreated subjects to better study the effectiveness and also the undesirable effects of Vaginal Filler and to guarantee scientifically valid and bias-free results.

INTERVENTIONS:
Device: Injections of a filler gel containing cross-linked hyaluronic acid — Vaginal Filler will be administered according to Investigator's judgment and Instruction For Use (IFU) to correct hypotrophy, improve the shape and increase the volume of the female external genital areas (labia majora). Vaginal Filler is a resorbable medical device available in packages containing 2 sterile pre-filled mono-use syringes of 1 ml with pre-assembled plunger rod and backstop, containing 25 mg/g cross-linked hyaluronic acid.
  The injection is performed by medical personnel at visit V0 in one or both sides of the superficial subcutaneous layer of the labia majora, along its longitudinal axis.The dosage to be used for the individual case is at the doctor's discretion. An anesthetic may be applied (lidocaine 2% injection only in the cannula access point) to the affected area before the IP injection.
  In order to maintain the results achieved, an eventual touch-up could be performed one months after the first treatment in the same areas of the first injection, at visit V2.
  Arms: Treatment Group (Vaginal Filler)

SUMMARY:
The overall aim of this research is to gather more information on the effectiveness of the Vaginal Filler medical device used in women to correct the thinning of the external genital tissue of the labia majora, re-proportioning its volume in relation to the labia minora and improving sexual function. It will also collect data about the safety and tolerability of Vaginal Filler.

The main question it aims to answer is:

• Does the treatment with Vaginal Filler medical device lead to an improvement of sexual functions in women with atrophy of female external genitalia (labia major)?

Researchers will compare subjects treated with Vaginal Filler medical device to untreated subjects to better study the effectiveness and also the undesirable effects of Vaginal Filler and to guarantee scientifically valid and bias-free results.

Participants will:

* receive the Vaginal Filler device via microinjections into the labia majora, if assigned to the Vaginal Filler treatment group;
* Attend the clinic for 6 scheduled visits: screening visit (V-1), baseline visit (V0) with the execution of the treatment and 4 subsequent follow-up visits (V1, V2, V3, V4) carried out 2 weeks, 1, 3 and 6 months after V0. The total duration of the study will be approximately 6 months;
* Keep a daily diary of any disorders, health problems or adverse events that may occur;
* Complete some questionnaires during the visits to the clinic.

DETAILED DESCRIPTION:
With the natural ageing process, the entire body is affected by structural and morphological physical changes, including the female external genitalia (vulva). These tend to wither and lose the characteristics of youthful age, compromising the sexual sphere and quality of life.

This phenomenon depends on the physiological hormonal changes typical of menopause, which inevitably lead to major aesthetic, physical and psychological changes.

The female genital apparatus, around the age of 40 to 50, changes not only due to advancing age but also due to the lack of oestrogen (the main female sex hormones), which progressively decreases until it disappears, leading to a progressive change in the structure of the vaginal and vulvar tissue.

The decrease in hyaluronic acid, elastic fibres, collagen, and the fatty layer results in a macroscopic loss of volume, noticeable skin laxity, and a change in the ratio between the labia majora and labia minora, which causes the latter to protrude more.

The reduced volume and change in the shape of the labia majora compromise their protective function of the internal structures, exposing the labia minora and vagina to microtrauma that contributes to certain menopausal symptoms such as dryness, burning, pain and itching of the innermost structures.

This condition, named vulvo-vaginal atrophy, is still little known, although it affects 1 in 2 post-menopausal women.

There are several approaches for the treatment of this condition. A wide range of surgical techniques is available for reducing the labia minora, mostly based on marginal excision or resection of the protruding parts of the labia minora.

Augmentation of the labia majora, on the other hand, is a relatively new technique for which there is currently no standardised approach and there are not many studies on it.

Aesthetic medicine can improve the appearance not only of the face and body but also of the intimate parts.

Currently, hyaluronic acid fillers are widely used for skin rejuvenation, and vulvar fillers can be used for both aesthetic and functional purposes.

Hyaluronic acid is a natural substance that is fundamental to the tissues of all mammals and is mainly found in the deepest part of the skin.

Its biological function, in addition to its structural function, plays an important role in wound healing, skin renewal and modulation of the immune response.

Hyaluronic acid injection in dermaesthetics is widely used with success, as it is considered safe due to the substance's complete reabsorbability and excellent tolerability, and provides excellent three-dimensional volume restoration of the treated area. In addition, the treatment is carried out on an outpatient basis.

The product that is the subject of this clinical study, Vaginal Filler, is a class III medical device already on the market, whose gel formulation combines different types of high and low molecular weight hyaluronic acid, which provide better stability and consistency and ensure long duration and permanence in the site of interest.

Moreover, the derivation of hyaluronic acid from bacterial and non-animal fermentation guarantees a sterile and high-quality product, preventing possible allergic reactions.

Vaginal Filler is intended for the treatment of atrophy and volume enhancement of the female external genital areas (labia majora).

The aesthetic result is very natural and long-lasting (up to 8-12 months), depending on individual characteristics (skin type, individual metabolism, anatomy, age) and lifestyle.

The primary objective of the study is to evaluate the efficacy of Vaginal Filler, used according to the intended indications, in correcting atrophy of the female external genitalia (labia majora), with re-proportioning of the ratio between the labia minora and labia majora and improvement of sexual function.

The secondary objectives of the study are to assess:

1. the impact of Vaginal Filler used to improve sexual function;
2. the performance of Vaginal Filler in improving the participant's quality of life;
3. the performance of Vaginal F iller in reducing the demand for labiaplasty of the labia minora, in the absence of actual hypertrophy
4. the performance of Vaginal Filler used for vulvar remodelling;
5. the performance of Vaginal Filler in alleviating the symptoms of vulvar atrophy and hypotrophy;
6. the intensity of the participant's pain following Vaginal Filler injection;
7. the satisfaction of the participant following the use of Vaginal Filler;
8. the safety of use and tolerability of Vaginal Filler.

The study plans to include 76 female subjects aged 40-65 years, who are affected by atrophy and/or hypotrophy (mild to severe) of the labia majora.

This research will contribute to the collection of data and the acquisition of new knowledge regarding the efficacy, safety of use and tolerability of Vaginal Filler and its application in aesthetic and functional gynaecology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Informed consent form (ICF) signed;
* Female aged 40-65 years;
* Atrophy and/or hypotrophy of labra majora requiring volume augmentation. Hypotrophy will be preoperatively staged in mild, moderate and severe considering both the adipose tissue and the cutaneous layer;
* Body Mass Index (BMI)<32 Kg/m2;
* Willingness to follow all study procedures, including attending all site visits, tests and examinations.

Exclusion Criteria:

* Allergy or controindications to device components;
* Allergy or controindications to anesthetic components;
* Previous surgery on external genitalia;
* Infectious or inflammatory processes close to the area of the procedure;
* History of vulvar cancer (including vulvar squamous papillomas) and/or previous regional radiotherapy;
* Active local herpes simplex or herpes zoster infection;
* Active herpes zoster infection in other sites;
* Active skin allergy including local dermatitis;
* Chronic pathological skin condition;
* Active mycosis and others bacterial infections;
* Immune system illnesses/disease;
* Known hypersensitivity to cheloids;
* Diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder);
* Problems with coagulation or anti-coagulating therapies in progress;
* Current treatment with substances which act on blood fluidity (eg. Aspirin, NSAIDs, Vitamin C), anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago), drugs able to influence the test results in the investigator opinion;
* Known drug and/or alcohol abuse;
* Mental incapacity that precludes adequate understanding or cooperation;
* Pregnancy or breastfeeding;
* COVID-19 vaccination within two month prior to study inclusion;
* Participation in another investigational study within 1 month prior to study inclusion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of the performance of Vaginal Filler in improving sexual functions. | At the end of the study (Visit V4) 6 months after enrolment.
  The Female Sexual Function Index (FSFI) will be used to evaluate the improvement of sexual functions at the end-of-study visit, comparing the results between the treatment and the control group. This questionnaire consists of 19 questions addressed to the patient, who can answer with a score from 0 or 1 (worst result) to 5 (best result).

SECONDARY OUTCOMES:
Evaluation of the performance of Vaginal Filler in improving sexual functions. | At V0 (Baseline visit day 0, before IP administration), V1 (2 weeks from V0), V2 (1 month from V0), V3 (3 months from V0) and V4 (6 months from V0).
  The Female Sexual Function Index (FSFI) will be used to evaluate the improvement of sexual functions at each study visit, comparing the results between the treatment and the control group. This questionnaire consists of 19 questions addressed to the patient, who can answer with a score from 0 or 1 (worst result) to 5 (best result). At baseline visit V0, the FSFI will be evaluated pre-injection; the pre-injection scores will be considered as baseline value.
Evaluation of the performance of Vaginal Filler in improving subjects' quality of life. | At V0 (Baseline visit day 0), V1 (2 weeks from V0), V2 (1 month from V0), V3 (3 months from V0) and V4 (6 months from V0).
  Subjects' Quality of Life (QoL) will be assessed at each study visit using the Perceived Stress Scale (PSS), comparing the results between the treatment and the control group. This questionnaire consists of 10 questions addressed to the patient, who can answer with a score from 0 (never) to 5 (usually).
Evaluation of the performance of Vaginal Filler in improving the shape and re-proportioning the ratio between labia minora and labia majora. | At V0 (Baseline visit day 0, before and after IP administration), V1 (2 weeks from V0), V2 (1 month from V0), V3 (3 months from V0) and V4 (6 months from V0).
  Labia minora hypertrophy classification will be performed using the S. Motakef Classification at each visit. Labial protrusion will be assessed measuring, with the help of tweezers and a ruler, the distance of the lateral edge of the labia minora from that of the labia majora. Three classes of labial protrusion could be identified: class I protrusion from 0 to 2 cm, class II , from 2 to 4 cm, and class III ,protrusion >4 cm. At V0, labial protrusion will be evaluated pre and post injection; the pre-injection score will be considered as baseline value.
Evaluation of the performance of Vaginal Filler for vulvar reshaping. | At V0 (Baseline visit day 0, before and after IP administration), V1 (2 weeks from V0), V2 (1 month from V0), V3 (3 months from V0) and V4 (6 months from V0).
  The change in the Global Aesthetic Improvement Scale (GAIS) between the treatment and the control group will be utilized to assess the performance of Vaginal Filler for vulvar reshaping. For evaluation of the GAIS, 2D photographs will be taken using an I-phone with standardized settings. Subjects should be photographed in frontal gynecological position and at 45° right and left and cranio-caudal orientation as well as in frontal upright position.
  The GAIS is a five-point scale for assessing global aesthetic improvement, where a score of 1 corresponds to the optimal cosmetic result and 5 to a worsening of appearance compared to the original condition.
  At V0, the GAIS will be evaluated pre and post injection; the pre-injection scores will be considered as baseline value. The GAIS will be completed independently by both the subjects and the physician investigators.
Evaluation of the performance of Vaginal Filler to alleviate the symptoms of vulvar atrophy and hypotrophy. | At V0 (Baseline visit day 0), V1 (2 weeks from V0), V2 (1 month from V0), V3 (3 months from V0) and V4 (6 months from V0).
  The Visual Analog Scale (VAS) will be used to assess the impact of Vaginal Filler on the symptoms of vulvar atrophy and hypotrophy at each visit. VAS is a straight horizontal line of fixed length (100 mm). The ends are defined as the extreme limits of the parameter to be measured (improvement of symptoms related to vulvar hypotrophy and atrophy) orientated from the left (0 - No improvement in symptoms) to the right (10 - Maximum improvement of symptoms). The patient should mark with a vertical line a point from 0 to 10 based on the perceived improvement in symptoms. The investigator will then measure the distance between the score 0 and the mark made by the patient with a 10-cm ruler and record the data in digits to one decimal place.
  The VAS score of the treatment group will be compared with the score of the control.
Evaluation of pain intensity after injection of Vaginal Filler. | At V0 (Baseline visit day 0, after IP administration)
  To evaluate pain intensity after injection of Vaginal Filler, a Numerical Rating Scale (NRS) will be used at baseline visit V0. Only patients in the treatment group will be asked to fill out the NRS, selecting a number from 0 to 10 indicating the degree of pain experienced after the injection (0 - No pain; 10 - The most intense pain imaginable).
  The NRS can be administered verbally soon after the injection and by telephone after the injection in the case the anesthetic will be used. In this case, the Investigator should wait until the effect of the anesthetic is resolved before asking the Subject the numerical value that best describes her pain intensity.
Evaluation of patient tolerance and satisfaction with Vaginal Filler treatment. | At End-Of-Study visit (V4) (6 months after the treatment).
  At End-Of-Study visit (V4), patience tolerance and overall satisfaction with Vaginal Filler treatment will be assessed by means of 5-point Likert Scale. Only patients in the treatment group will be asked to fill out the Likert Scale, selecting a number from 1 to 5 that better corresponds to the degree of satisfaction about the treatment (0 - Not satisfied at all; 5 - Totally satisfied).
Safety monitoring through vulva examination. | From V-1 (Screening visit Week -1) to V4 (End of Study) at 6 months.
  Safety data including examination of the vulva and vital signs of the patient will be collected at each visit.
  During the screening phase (V-1), a gynecological examination will be performed to assess the presence of vulvar reddening, small fissures, fibrous whitish areas, ecchymosis and lacerations. Any abnormality identified at screening should be recorded on the General Medical History of CRF as Baseline Conditions. At subsequent visits (or as clinically indicated), limited, symptom-directed vulvar examinations should be performed. Changes from baseline abnormalities should be recorded in patient notes. New or worsened abnormalities after screening should be recorded as adverse events if appropriate.
Assessment of device deficiency/incidents. | At baseline visit V0 and eventually at visit V2 (in case of touch-up one month after the first treatment).
  Device deficiency/incident information will be collected by the investigator or its delegates on the CRF's.
Collection of any adverse events and serious adverse events. | From baseline visit (V0) to the end of the study (V4) at 6 months.
  Adverse event (AE) and adverse device effect information will be collected throughout the study. The event, date of onset, severity, duration, and relationship to the device will be recorded. Any AE will be monitored until it is adequately resolved or explained. All subjects will be also requested to report in a diary any adverse effect, in order to allow the Investigator to take the best decision to ensure the safety and well-being of trial subjects. During scheduled visits, patients will be properly interviewed by the medical staff to evaluate any adverse event. All AEs reported by the subject, observed by the Investigator, or documented in medical records will be recorded in the CRF, whether believed by the Investigator to be related or unrelated to the investigational device. Starting with the study enrollment, any new event/experience that was not present at baseline, or worsening of an event present at baseline, is considered an AE.
Assessment of concomitant medications. | From screening visit (V-1) to the end of the study (V4) at 6 months.
  All concomitant medications should be registered by the investigator on the appropriate page in the electronic case report form (eCRF) with the dosage and the medication (active substance).
  During the study, subjects will also be asked to record side effects and concomitant medications in a diary that will be dispensed at visit V0. At each scheduled visit, the investigator or delegates will properly interview the patients and check the diary to evaluate any concomitant medication.
Safety monitoring through vital signs by Blood Pressure. | From V-1 (Screening visit Week -1) to V4 (End of Study) at 6 months.
  Safety data including examination of the vulva and vital signs of the patient will be collected at each visit. Blood Pressure (systolic and diastolic pressures in mmHg) will be recorded for each patient using a sphygmomanometer.
Safety monitoring through vital signs by Heart Rate. | From V-1 (Screening visit Week -1) to V4 (End of Study) at 6 months.
  Safety data including examination of the vulva and vital signs of the patient will be collected at each visit. Heart Rate (beats/min) will be recorded for each patient using a sphygmomanometer.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele di Milano, Milan, Milan, Italy